CLINICAL TRIAL: NCT02682771
Title: Effects of Positive Airway Pressure and Incentive With Load Inspiratory on Lung Function and Respiratory Muscle in Post-bariatric Surgery - a Randomized and Blind Clinical Trial
Brief Title: Positive Airway Pressure Versus Breathing Exercises With Load Inspiratory in Patients Undergoing Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Responsible Party: Principal Investigator, Eli Maria Pazzianotto Forti, Principal Investigator, Universidade Metodista de Piracicaba
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: UMetodistaPiracicaba
Record Dates: First submitted 2016-01-22; First posted 2016-02-15 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Inadequate or Impaired Respiratory Function
Keywords: gastroplasty, breathing exercices, positive pressure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Active Comparator): Individuals were treated with Conventional Respiratory Physiotherapy (CRP), twice in immediate postoperative day and three times in first postoperative day.
  Interventions: Procedure: Conventional Respiratory Physiotherapy (CRP)
- Bilevel positive airway pressure (Experimental): Individuals were treated with positive pressure, in the BIPAP mode (bilevel positive airway pressure, with inspiratory pressure:12 cmH20 and expiratory pressure: 8 cmH20) twice in the immediate postoperative day and three times in first postoperative day, in sessions 1 hour each
  Interventions: Device: Bilevel positive airway pressure; Procedure: Conventional Respiratory Physiotherapy (CRP)
- Load inspiratory breathing exercises (Experimental): Individuals were treat with PowerBreathe, a device for inspiratory muscle, with 40% maximal inspiratory pressure, measured at preoperative, twice in the immediate postoperative day and three times in first postoperative day, in sessions 1 hour each.
  Interventions: Device: PowerBreathe; Procedure: Conventional Respiratory Physiotherapy (CRP)

INTERVENTIONS:
Device: Bilevel positive airway pressure — The use of positive airway pressure airway seeking in the prevention or treatment of hypoxic respiratory failure, improved arterial oxygenation, restoration or maintenance of lung volume reduction and atelectasis, decrease the work of breathing, decreased dyspnea index and increased residual volume
  Arms: Bilevel positive airway pressure
Device: PowerBreathe — Exercises with inspiratory load has the aim to trainning inspiratory muscle in strength and endurance, thus, could help to prevent postoperative complications.
  Arms: Load inspiratory breathing exercises
Procedure: Conventional Respiratory Physiotherapy (CRP) — CRP consisted of diaphragmatic respiratory exercises, deep inhalation exercises, inhalations fragmented two to three times and respiratory exercises associated with shoulder flexion movements and extension of the upper limbs. One series of 10 repetitions was carried out for each exercise. Walking sessions and preventive exercises for deep vein thrombosis were carried out

SUMMARY:
Obesity, due to excess fat in the thoracoabdominal region, can promote changes in respiratory function and lung function, leading to reduction in lung volume and capacity. Such dysfunctions are worsen after bariatric surgery to be associated with factors inherent to this procedure. The objective of this study was to evaluate and compare the effects of the application of bilevel positive airway pressure and exercises with inspiratory pressure with linear load in thoracoabdominal mobility, pulmonary function, inspiratory muscle strength, respiratory muscle strength and prevalence of pulmonary complications after bariatric surgery.

DETAILED DESCRIPTION:
This is a clinical trial, randomized, blinded, in which 60 volunteers, after evaluation preoperatively, consisting of: cirtometry to measure thoracoabdominal mobility, spirometry for measures of lung function, nasal inspiratory pressure to inspiratory muscle strength and endurance incremental test for evaluation of respiratory muscle strength, were randomized and allocated into three groups, with 20 volunteers each. The interventions were performed in the immediate postoperative period and the first day after surgery. The first group, called the control group received care by Conventional Respiratory Physiotherapy (CRP), consisting of breathing exercises, incentive spirometer and ambulation. The second group, called Positive Pressure Group received two-level positive airway pressure for one hour, addition of CRP. The third group, called Load Inspiratory Group held exercises with inspiratory pressure with linear load, linked also to the CRP. Treatments were applied twice in the immediate postoperative period and shortly after returning to the ward and after 4 hours of the initial treatment and three times a day on the first day after surgery. On discharge, the second day after surgery, the volunteers performed chest x-ray and underwent the same evaluations performed preoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Submitted to Roux-en-Y type gastric bypass by laparotomy
* Normal preoperative pulmonary function and chest x-ray

Exclusion Criteria:

* Hemodynamic instability
* Hospital Stay longer than three days
* Presence of postoperative complications
* Smoking
* Respiratory chronic diseases

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pulmonary function | up to 2 days after surgery
  Spirometry was carried out according to the guidelines of the American Thoracic Society (ATS) and European Respiratory Society (ERS) (2005). Three types of maneuver were used in order to evaluate the lumg volumes and flows: slow vital capacity, forced vital capacity and maximum voluntary ventilation. The maneuvers were carried out until three acceptable and reproducible curves were obtained, not exceeding more than eight attemps. The values extracted from each maneuver were selected according to Pereira (2002) and the predicted values calculated using the equation proposed by Pereira et al (1992( for Brazilians.

SECONDARY OUTCOMES:
Thoracoabdominal mobility | up to 2 days after surgery
  The measurement of thoracoabdominal mobility was performed by using a tape scaled in centimeters. In the standing position, the measurement were made at levels axillary, xiphoid and abdominal during rest and at maximal inspiration and maximal expiration. At each level, the measurements were performed three times. It computed the highest value of inspiration and lowest of expiration. The absolute difference between these values was considered the thoracoabdominal mobility.
Evaluation of inspiratory muscle endurance | up to 2 days after surgery
  The endurance test was performed using the PowerBreathe K3. An incremental test was performed, initiating at 30% of maximal inspiratory pressure for 30 respiratory cycles and then, added 10 cmH20 for each respiratory cycle. The test was finished when the individual was unabled to promote inspiratory effort.
Evaluation of muscle strength inspiratory | up to 2 days after surgery
  The Sniff is an alternative non-invasive technique for the assessment of inspiratory muscle strength by sniff nasal inspiratory pressure (PNSN). The measurement is performed using a peak pressure generated by nasal nostril during a maximal sniff from functional residual capacity

CONTACTS AND LOCATIONS:
Overall Officials: Eli Maria Pazzianotto-Forti, PhD, Principal Investigator — Universidade Metodista de Piracicaba
Locations (1):
- Universidade Metodista de Piracicaba, Piracicaba, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No